CLINICAL TRIAL: NCT05144373
Title: Role of Early Motor Experience in Infants With Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jianhua Wu, Professor, Georgia State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: H21604; 1R21HD105879-01 (NIH); 352307 (Other: National Institutes of Health)
Record Dates: First submitted 2021-10-05; First posted 2021-12-03 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Intervention Model Description: We will recruit 45 infants with DS from the greater Atlanta area and beyond. There will be three groups: (a) gross motor (GM) group (n=15), entering the study at about 10 months of age; (b) gross motor plus fine motor (GM+FM) group (n=15), entering the study at about 10 months; and (c) control group (n=15), entering the study at about 20 months. The GM group will receive a home-based, parent-guided practice of treadmill stepping from 10 months of age until walking onset. The GM+FM group will receive both treadmill intervention from 10 months of age until walking onset as well as fine motor experience in practice of grasping using "sticky mittens" from 10 months of age for about five months. The control group will not receive an intervention.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gross motor intervention (Experimental): Participants will receive a home-based, parent-administered body-weight supported treadmill intervention from about 10 months of age until walking onset.
  Interventions: Behavioral: Gross motor intervention, gross and fine motor intervention
- Gross and fine motor intervention (Experimental): Besides the body-weight supported treadmill intervention as illustrated above, participants will receive additional fine motor intervention using "sticky mittens" from about 10 months of age for five months.
  Interventions: Behavioral: Gross motor intervention, gross and fine motor intervention
- Control (No Intervention): Participants will not receive specific intervention.

INTERVENTIONS:
Behavioral: Gross motor intervention, gross and fine motor intervention — For gross motor intervention, participants will receive a home-based, parent-administered body-weight supported treadmill intervention from about 10 months of age until walking onset.
  For gross and fine motor intervention, participants will receive the same treadmill intervention as illustrated above. In addition, participants will receive a fine motor intervention with practice of reaching and grasping using "sticky mittens" from about 10 months of age for five months.
  Arms: Gross and fine motor intervention; Gross motor intervention

SUMMARY:
Infants with Down syndrome show significant delays and weaknesses in motor, cognitive, and language development compared to typically developing infants. This project aims to examine the developmental cascade effects of specific gross and fine motor experience on motor, cognitive and language development in infants with Down syndrome. We propose that both gross and fine motor experience will facilitate cognitive and language development in infants with Down syndrome, and particularly, fine motor experience will help advance gesture and early words production.

DETAILED DESCRIPTION:
Down syndrome (DS) is the most common genetic condition and causes significant development delays and weaknesses in the motor, cognitive, and language domains. It is important to study these co-occurring developmental challenges and develop effective intervention strategies for positive learning outcomes in multiple domains simultaneously. It was found that motor development is closely associated with cognitive and language development in typically developing infants and advances in motor development have developmental cascade effects on other domains. However, this interrelation has not been studied in infants with DS. Our prior work has shown that gross motor experience through body-weight-supported treadmill stepping leads to an earlier onset of walking and improves subsequent locomotor ability in infants with DS. However, we do not yet know the extent to which this motor experience advances cognitive and language development in infants with DS. Research also suggests that grasping, a major fine motor skill emerging in infancy, provides the needed scaffolding for subsequent gesture and speech production. However, research on grasping and its potential effects on other domains in infants with DS remains scarce. The objectives of this proposal are to understand: the role of (a) specific gross motor experience and (b) specific fine motor experience on the motor, cognitive and language development of infants with DS. Our central hypothesis is that motor (both gross and fine) experience will help advance cognitive and language development in infants with DS. We will recruit 45 infants with DS from the greater Atlanta area and beyond. There will be three groups: (a) gross motor (GM) group (n=15), entering the study at about 10 months of age; (b) gross motor plus fine motor (GM+FM) group (n=15), entering the study at about 10 months; and (c) control group (n=15), entering the study at about 20 months. Aim 1: Determine the effects of gross motor experience on cognitive and language development in infants with DS, comparing the GM and control groups. Only the GM group will receive a home-based, parent-guided practice of treadmill stepping from 10 months of age (T1) until onset of walking. We hypothesize that the GM group will show higher Bayley scores and better gesture and word production at termination of the GM intervention (T3) and five months thereafter (T4) than the control group. Aim 2: Determine the effects of fine motor experience on cognitive and language development in infants with DS who receive the GM intervention, particularly in gesture and word production, comparing the GM and GM+FM groups. Only the GM+FM group will receive fine motor experience in practice of grasping using "sticky mittens" from 10 months of age for about five months. We hypothesize that the GM+FM group will show further improvements in motor, cognitive and language domains, particularly in gesture and word production, than the GM group at termination of the FM intervention (T2) and again at T3 and T4. Our study will gain an in-depth understanding of the cascading effects of motor experience on cognitive and language development and lay the groundwork for future clinical trials in infants with DS.

ELIGIBILITY:
Inclusion Criteria:

* An appropriate age range of 7-36 months
* A diagnosis of Down syndrome.

Exclusion Criteria:

* The presence of seizure disorders
* Non-correctable vision, hearing and heart problems
* Any other severe medical conditions that may prevent the infant from participating in this study

Ages: 7 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Bayley cognitive scores | 10 months for GM and GM+FM groups
  The Bayley Scale of Infant and Toddler Development cognitive composite scores
Bayley cognitive scores | 15 months for GM and GM+FM groups
  The Bayley Scale of Infant and Toddler Development cognitive composite scores
Bayley cognitive scores | 20 months for all three groups
  The Bayley Scale of Infant and Toddler Development cognitive composite scores
Bayley cognitive scores | 25 months for all three groups
  The Bayley Scale of Infant and Toddler Development cognitive composite scores
Bayley language scores | 10 months for GM and GM+FM groups
  The Bayley Scale of Infant and Toddler Development language composite scores
Bayley language scores | 15 months for GM and GM+FM groups
  The Bayley Scale of Infant and Toddler Development language composite scores
Bayley language scores | 20 months for all three groups
  The Bayley Scale of Infant and Toddler Development language composite scores
Bayley language scores | 25 months for all three groups
  The Bayley Scale of Infant and Toddler Development language composite scores
Gesture production | 10 months for GM and GM+FM groups
  It measures the type, frequency, and quality of gestures that the infant produces during infant-parent interaction
Gesture production | 15 months for GM and GM+FM groups
  It measures the type, frequency, and quality of gestures that the infant produces during infant-parent interaction
Gesture production | 20 months for all three groups
  It measures the type, frequency, and quality of gestures that the infant produces during infant-parent interaction
Gesture production | 25 months for all three groups
  It measures the type, frequency, and quality of gestures that the infant produces during infant-parent interaction

SECONDARY OUTCOMES:
Bayley motor scores | 10 months for GM and GM+FM groups
  The Bayley Scale of Infant and Toddler Development motor composite scores
Bayley motor scores | 15 months for GM and GM+FM groups
  The Bayley Scale of Infant and Toddler Development motor composite scores
Bayley motor scores | 20 months for all three groups
  The Bayley Scale of Infant and Toddler Development motor composite scores
Bayley motor scores | 25 months for all three groups
  The Bayley Scale of Infant and Toddler Development motor composite scores

CONTACTS AND LOCATIONS:
Locations (1):
- Biomechanics lab, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
We will upload the data to the National Institutes of Health INCLUDE data coordination center (DCC). We will share the de-identified data including demographics, diagnosis, and motor, cognitive, and language developmental profile. We will also share the video data including the captured motion data and the footage of parent-child interaction.
Supporting Information: Study Protocol, ICF
Time Frame: We will deposit the de-identified data and video data into the National Institutes of Health INCLUDE data coordinating center (DCC) as soon as possible but no later than within one year of the completion of the funded project period for the parent award or upon acceptance of the data for publication, or public disclosure of a submitted patent application, whichever is earlier.